CLINICAL TRIAL: NCT01109095
Title: Administration of HER2 Chimeric Antigen Receptor Expressing CMV-Specific Cytotoxic T Cells Ins Patients With Glioblastoma Multiforme (HERT-GBM)
Brief Title: CMV-specific Cytotoxic T Lymphocytes Expressing CAR Targeting HER2 in Patients With GBM
Acronym: HERT-GBM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Nabil Ahmed, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-24487 - HERT GBM
Record Dates: First submitted 2010-04-13; First posted 2010-04-22 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Glioblastoma Multiforme (GBM)
Keywords: Glioblastoma Multiforme (GBM); HER2; CMV; Brain Cancer; Autologous HER2.CAR CMV-specific cytotoxic CTL; CMV-specific cytotoxic CTL
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HER.CAR CMV-specific CTLs (Experimental): Subject will be assigned a dose level at study entry.
  Interventions: Biological: HER.CAR CMV-specific CTLs

INTERVENTIONS:
Biological: HER.CAR CMV-specific CTLs — HER2.CAR CMV-specific CTLs will be given by intravenous injection over 1-10 minutes through either a peripheral or a central line with a minimum 20g cannula. The patient will get one of the following doses:
  * 1 x 10^6/m^2
  * 3 x 10^6/m^2
  * 1 x 10^7/m^2
  * 3 x 10^7/m^2
  * 1 x 10^8/m^2

SUMMARY:
This study is for patients that have a type of brain cancer called glioblastoma multiforme (GBM).

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise, but have not been strong enough to cure most patients.

The antibody used in this study is called anti-HER2 (Human Epidermal Growth Factor Receptor 2). This antibody sticks to GBM cells because of a substance on the outside of these cells called HER2. Up to 80% of GBMs are positive for HER2. HER2 antibodies have been used to treat people with HER2-positive cancers. For this study, the HER2 antibody has been changed so that instead of floating free in the blood it is now attached to T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These chimeric receptor-T cells seem to be able to kill tumors like GBM, but they don't last very long and so their chances of fighting the cancer are limited. Therefore, developing ways to prolong the life of these T cells should help them fight cancer.

We found that T cells work better if we also attach a protein called CD28 to the HER2 chimeric receptor (HER2-CAR). In this study we placed this HER2-CAR into T cells that were pre-selected for their ability to recognize Cytomegalovirus (CMV). This virus exists in most people. These CMV-specific cytotoxic T cells (CMV-T cells) will be more active since they will react to the virus as well as to tumor cells. These HER2-CD28 CMV-T cells are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to find the largest safe dose of HER2-CD28 CMV-T cells, to learn what the side effects are, and to see whether this therapy might help patients with GBM.

DETAILED DESCRIPTION:
When the patient enrolls on this study, they will be assigned to a dose of HER2-CAR CMV-T cells.

The patient will be given a single injection of cells into the vein through an IV line at the assigned dose. The injection will take between 1 and 10 minutes. The patient will be followed in the clinic after the injection for 1 to 4 hours. If later the subject seems to be experiencing a benefit (confirmed by radiological studies, physical exam and/or symptoms), s/he may be able to receive up to six additional doses of the T cells if they wish. These additional infusions would be at least 6 to 12 weeks apart and at the same dose level received the first time.

Medical tests before treatment--

Before being treated, the patient will receive a series of standard medical tests as follows: Physical exam, Blood tests to measure blood cells, kidney and liver function, Routine heart function tests (Echocardiogram),Measurements of the tumor by routine imaging studies

Medical tests during and after treatment--

The patient will receive standard medical tests when getting the infusions and after:Physical exams, Blood tests to measure blood cells, kidney and liver function, Routine heart function tests (Echocardiogram) at 6 weeks after the infusion, Measurements of the tumor by routine imaging studies 6 weeks after the infusion

To learn more about the way the HER2-CAR CMV-T cells are working and how long they last in the body, blood will be taken on the day of the T-cell infusion, before, 1 hour and 4 hours after the T-cell infusion, 1, 2, 4 and 6 weeks after the T-cell infusion and every 3 months for 1 year, every 6 months for 4 years, then yearly for a total of 15 years.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histopathological verification of glioblastoma multiforme (GBM: WHO grade IV) with recurrent or progressive disease after front line therapy.
* HER2 positive GBM
* CMV seropositive
* Normal ECHO (Left ventricular ejection fraction (LVEF) has to be with in normal, institutional limits)
* Life expectancy 6 weeks or greater
* Karnofsky/Lansky score 50 or greater
* Patient or parent/guardian capable of providing informed consent
* Bilirubin 3x or less than normal, AST 5x or less than normal, creatinine 2x normal or less for age and Hgb 9.0 g/dl or more; WBC greater than 2,000/ul; ANC greater than 1,000/ul; platelets greater than 100,000/ul
* Pulse oximetry 90% or more on room air
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the CTL infusion. The male partner should use a condom.
* Available autologous HER2.CAR-transduced CMV-specific cytotoxic T lymphocytes with 15% or greater expression of HER2.CAR determined by flow-cytometry and killing of HER2-positive targets 20% or more in cytotoxicity assay.
* Recovered from the acute toxic effects of all prior chemotherapy at least 4 weeks before entering this study. One exception is Temozolomide(TMZ), an alkylation agent used as a radiosensitizer and adjuvant chemotherapeutic agent for GBM. Due to the extremely short half life of TMZ, patients will be allowed to continue receiving it up to two days prior to cell infusion and cannot restart until six weeks after the infusion.

EXCLUSION CRITERIA:

* Severe intercurrent infection
* Known HIV positivity
* Pregnant or lactating
* History of hypersensitivity reactions to murine protein-containing products

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicity after CTL infusion | 6 weeks
  To evaluate the safety of escalating doses of autologous CMV-specific cytotoxic T-lymphocytes (CTL) genetically modified to express chimeric antigen receptors (CAR) targeting the HER2 molecule in patients with HER2-positive Glioblastoma multiforme (GBM: WHO grade IV), who have recurrent or progressive disease after front line therapy.

SECONDARY OUTCOMES:
Decrease in tumor after the CTL infusion | 6 weeks
  To evaluate the effects of gene modified CTL on measurable disease.
Area under the growth curves (AUC) over time for T cell frequencies. | 15 years
  To measure the survival and function of gene modified CTL in vivo.
Impact of gene modified CTL on CMV-specific T lymphocyte immune response | 15 years
  Immune function assays including ELISPOT or CTLp assays and cytotoxicity assays to look at specificity of response will be done in patients on whom the appropriate reagents are available

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Ahmed, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Badhiwala J, Decker WK, Berens ME, Bhardwaj RD. Clinical trials in cellular immunotherapy for brain/CNS tumors. Expert Rev Neurother. 2013 Apr;13(4):405-24. doi: 10.1586/ern.13.23. PMID 23545055